CLINICAL TRIAL: NCT03494855
Title: Reducing Scan Times and Improving Care Through Quantitative Imaging: Evaluating the Efficacy of SyMRI in Clinical Pediatric Populations
Brief Title: Evaluating the Efficacy of SyMRI in Clinical Pediatric Populations
Acronym: SyMRI
Status: Terminated | Type: Observational
Why Stopped: Patient accrual is slow and software renewal is costly and beyond our allocated fund for this study.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Manohar Shroff, Chief Radiologist, The Hospital for Sick Children
Other Study IDs: 1000048815
Record Dates: First submitted 2018-01-17; First posted 2018-04-11 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Brain Injuries; Brain Development Abnormality; Brain Pathology
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Neonates: <1 month of age SyMRI software used for brain imaging and radiological interpretation
  Interventions: Device: SyMRI Software
- Infants: 1mth - 2 years of age SyMRI software used for brain imaging and radiological interpretation
  Interventions: Device: SyMRI Software
- Adolescents: 2 - 12 years of age SyMRI software used for brain imaging and radiological interpretation
  Interventions: Device: SyMRI Software
- Teenagers: 13-18 years of age SyMRI software used for brain imaging and radiological interpretation
  Interventions: Device: SyMRI Software
- Healthy Adults: Preliminary Evaluation SyMRI software used for brain imaging and radiological interpretation
  Interventions: Device: SyMRI Software

INTERVENTIONS:
Device: SyMRI Software — The MDME sequence aims to provide whole absolute quantification of T1, T2, PD and B1 inhomogeneity in 5 minutes at typical clinical resolution (0.8 x 0.8 x 5mm). SyMRI software then allows a user to synthesize any almost image contrast (T1, T2, PD, FLAIR, IR, DIR, etc) by adjusting imaging parameters after the fact.

SUMMARY:
Synthetic MR Technologies has created a quantified imaging solution - SyMRI - to enable radiologists to acquire quantified images and always obtain the best contrast images. This study represents an attempt to assess the clinical utility of this software.

DETAILED DESCRIPTION:
Typical magnetic resonance imaging (MRI) involves taking many images called 'contrasts' to look at the body in different ways. Standard scan settings are usually good enough for a radiologist to review. The best settings often change with the age of the patient and their health, and are time consuming to determine. Quantified imaging is an alternative to contrast-based imaging which explicitly measures tissue properties and can be used to create almost any contrast. This method of imaging has been held back by a lack of the right software. Synthetic MR Technologies has created a quantified imaging solution - SyMRI - to enable radiologists to acquire quantified images and always obtain the best contrast images.

The objective of this study is to evaluate SyMRI in a pediatric population to determine if Sickkids would be interested in purchasing this product / support Health Canada approval. Specifically, the investigators are interested in determining if SyMRI is clinically useful:

* Is synthetic imaging quality comparable / better than conventional imaging?

  * Qualitative - Are radiologists more confident using synthetic MR vs conventional
  * Quantitative - Signal-to-noise (SNR) and Contrast-to-noise (CNR)
* To what extent can total exam times be reduced?
* Is the software user friendly and would investigators use it?

ELIGIBILITY:
Inclusion Criteria:

* Any stable patient undergoing clinical MRI of the brain is eligible for this study.
* Research patients undergoing research MRI of the brain for another study will be eligible.

Exclusion Criteria:

* Only those patients where an additional 10 minutes of MR imaging would not be advisable (ie. unstable, implants) or possible (due to scheduling constraints) will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Preliminary evaluation - 6 adult volunteers (>18 years of age)
  2. Clinical Evaluation
  i) 25 neonates (<1 month of age) ii) 25 infants (1mth - 2 years of age) iii) 25 adolescents (2 - 12 years of age) iv) 25 teenagers (13-18 years of age)
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Quality relative to conventional imaging | Through study completion, an average of 1 year
  Radiologist compares qualitative diagnostic quality of SyMRI imaging against Conventional Imaging.
  Measure - Poorer, Equal, Better

SECONDARY OUTCOMES:
Scan time for SyMRI vs Conventional MR | Through study completion, an average of 1 year
  Compare acquisition time for SyMRI scans vs Conventional MR Measure - Minutes:Seconds

CONTACTS AND LOCATIONS:
Overall Officials: Manohar Shroff, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03494855/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03494855/SAP_001.pdf